CLINICAL TRIAL: NCT01302197
Title: Muscle Atrophy, Physical Performance and Glucose Tolerance Post Stroke
Status: Active, not recruiting | Type: Observational
Sponsor: Baltimore VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alice S. Ryan, PhD, Professor of Medicine, Baltimore VA Medical Center
Other Study IDs: HP-00042905
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: Stroke; Body Composition; Glucose Tolerance
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be analyzed for metabolic biomarkers. Muscle tissue is collected for measurements of muscle phenotype. A urine pregnancy test is performed in women of child bearing age before CT imaging to exclude pregnant women due to the risk to an unborn fetus.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — longitudinal follow-up after stroke

SUMMARY:
Stroke, a leading cause of disability in the aging population, increases the risk for diabetes, subsequent stroke recurrence, and cardiovascular disease complications. The downsizing of private and federal health care resources, along with the anticipated increase in stroke rates as our population ages, mandate that alternative strategies be developed to reduce the public health burden of stroke. This pilot study may facilitate our knowledge of the timing of paretic leg muscle atrophy, fiber type shift, and the progression of worsening of glucose tolerance after stroke. Knowledge of the skeletal muscle changes occurring in the sub-acute stroke period is essential to create new guidelines incorporating exercise rehabilitation, much like cardiac rehabilitation, in order to facilitate and improve the health care of veteran stroke survivors.

DETAILED DESCRIPTION:
The vast majority of cerebrovascular accidents are reported in persons older than 55 years of age and occur in over 780,000 persons each year in the U.S. As our adult population ages, the number of strokes in the United States is anticipated to double, reaching nearly 1.5 million annually by the year 2050. Following stroke, patients remain at continued high risk for recurrent stroke with almost a third of them suffering recurrent stroke within 5 years, even despite optimal medical management. Age and cardiac disease are among the most important longitudinal predictors of cardiovascular health outcomes and survival after stroke. Notably, 75% of chronic stroke survivors have residual disability emphasizing the need for rehabilitation strategies.

Knowledge of the skeletal muscle changes that occur in the early phases after stroke is essential to create new guidelines which incorporate exercise rehabilitation, much like cardiac rehabilitation, in order to facilitate and improve the health care of stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 21 years of age or older
* BMI between 20-50 kg/m2
* Presenting within a month after stroke onset with residual hemiparetic deficit
* Patients must have adequate language and neurocognitive function to participate in testing and give adequate informed consent

Exclusion Criteria:

* Patients deemed too disabled to participate in physical therapy, or patients with minimal deficits, or patients who fully recovered after their stroke, in which physical therapy is not necessary
* Unstable angina, CHF, severe PAD
* Dementia or untreated major depression
* Severe receptive or global aphasia
* Heavy alcohol use defined by greater than 3 oz. liquor, 12 oz of wine or 32 oz of beer daily
* Muscle biopsy Exclusion Criteria:

  * anti-coagulation therapy with heparin, warfarin, or lovenox (anti-platelet therapy is permitted)
  * bleeding disorder
  * allergy to lidocaine

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Stroke
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-04-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in body composition | change in muscle mass from baseline to 3 months
  Muscle mass

SECONDARY OUTCOMES:
Change in glucose | change in glucose from baseline to 3 months
  glucose levels
Change in physical function | change in walk distance from baseline to 3 months
  walk distance

CONTACTS AND LOCATIONS:
Overall Officials: Alice S Ryan, Ph.D., Principal Investigator — University of Maryland School of Medicine, Baltimore VA Research Service
Locations (3):
- United States (3):
  - University of Maryland Medical System, Baltimore, Maryland
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - Kernan Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No